CLINICAL TRIAL: NCT05363722
Title: A Randomized, Open-label, Multicenter Phase Ib Clinical Study to Observe the Effectiveness and Safety of Different Doses of IBI310,Bevacizumab Combined With Sintilimab in the First-line Treatment of Advanced Hepatocellular Carcinoma
Brief Title: A Clinical Study to Observe the Effectiveness and Safety of IBI310, Bevacizumab Combined With Sintilimab in the Treatment of Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310Y001
Record Dates: First submitted 2022-04-14; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A（IBI310 0.5mg/kg） (Experimental): IBI310 0.5mg/kg IV d1 Q6W, sintilimab 200mg IV d1 Q3W, combined with bevacizumab 15mg/kg IV d1，Q3W
  Interventions: Drug: IBI310（0.5mg/kg）; Drug: sintilimab; Drug: bevacizumab
- Arm B（IBI310 0.3mg/kg） (Experimental): IBI310 0.3mg/kg IV d1 Q6W, sintilimab 200mg IV d1 Q3W, combined with bevacizumab 15mg/kg IV d1，Q3W
  Interventions: Drug: IBI310（0.3mg/kg）; Drug: sintilimab; Drug: bevacizumab

INTERVENTIONS:
Drug: IBI310（0.5mg/kg） — IBI310 0.5mg/kg IV d1 Q6W
  Arms: Arm A（IBI310 0.5mg/kg）
Drug: IBI310（0.3mg/kg） — IBI310 0.3mg/kg IV d1 Q6W
  Arms: Arm B（IBI310 0.3mg/kg）
Drug: sintilimab — sintilimab 200 mg IV d1 Q3W
Drug: bevacizumab — bevacizumab 15 mg/kg IV d1，Q3W

SUMMARY:
This is a randomized, open-label, multicenter Phase Ib study to evaluate the effectiveness and safety of different doses of IBI310, bevacizumab combined with sintilimab in patients with locally advanced or metastatic HCC who have not previously received systemic therapy, are unsuitable for radical surgical resection or local treatment, or have progressive disease after surgical resection or local treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed hepatocellular carcinoma, or meeting the clinical diagnostic criteria for hepatocellular carcinoma ;
2. Aged ≥18 years,≤75 years;
3. ECOG performance status score of 0 or 1 point;
4. Barcelona Clinic Liver Cancer (BCLC) stage C, or Stage B not suitable for radical surgery and/or local treatment;
5. No systemic antitumor treatment for hepatocellular carcinoma before the first administration;
6. At least 1 measurable lesion according to the Response Evaluation Criteria in Solid Tumors Version 1.1(RECIST V1.1), or measurable lesion with definite progression after local treatment (based on RECIST V1.1 criteria);
7. Child-Pugh Class A or B(≤7);
8. Adequate organ and bone marrow function.
9. Expected life time is over 12 weeks.
10. Take effective contraceptive measures
11. Willing to attend the study and having given the ICF

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, mixed cholangiocarcinoma and HCC
2. History of hepatic encephalopathy or liver transplantation
3. Pleural, ascites, and pericardial effusion with clinical symptoms requiring drainage
4. HBV-DNA>2000 IU/ML or 10^4 copies/ml；Untreated positive HCV-RNA；HbsAg and anti-HCV antibody were both positive
5. History of GI bleeding within 6 months, or severe (G3) varices at endoscopy within 3 months
6. Arteriovenous embolism within 6 months
7. The tumor thrombus involved both main and branch portal veins, main portal veins and mesenteric veins or inferior vena cava.
8. Antiplatelet drugs were administered for 10 days for therapeutic purposes 2 weeks before administration
9. Uncontrolled hypertension
10. Unrecovered AE（>CTCAE grade 1） due to previous treatment
11. Heart failure (NYHA Classification III-IV), or poorly controlled arrhythmias
12. History of gastrointestinal perforation, fistula, intestinal obstruction, extensive bowel resection, Crohn's disease, ulcerative colitis, or chronic diarrhea
13. With lung fibrosis, interstitial lung disease, pneumoconiosis, drug-associated pneumonia and serious impairment in lung function
14. Active tuberculosis
15. Infected with HIV or syphilis
16. Severe infections that are active or clinically poorly controlled
17. Use of immunosuppressive drugs within 4 weeks prior to initial dosing
18. Receipt of live attenuated vaccine within 4 weeks prior to randomization
19. Significant traumatic injury or major surgical procedure within 28 days prior to randomization
20. Other conditions that the investigator judged inappropriate for inclusion
21. Prior immunotherapy or targeted therapy
22. Treatment of Traditional Chinese medicine with anti-tumor indications or drugs with immunomodulatory effects whitin 2 weeks
23. Pregnant or breast-feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | The proportion of patients with complete response or partial response, through study completion, an average of 3 years
  efficacy

SECONDARY OUTCOMES:
Duration of Response（DOR）according to RECIST V1.1 criteria | From date of randomization until the date of first documented progression, up to 48 months
  efficacy
Duration of Response（DOR）according to mRECIST criteria | From date of randomization until the date of first documented progression, up to 48 months
  efficacy
Disease Control Rate（DCR） according to RECIST V1.1 criteria | The percentage of patients whose therapeutic intervention has led to a complete response, partial response, or stable disease, through study completion, an average of 3 years
  efficacy
Disease Control Rate（DCR） according to mRECIST criteria | The percentage of patients whose therapeutic intervention has led to a complete response, partial response, or stable disease, through study completion, an average of 3 years
  efficacy
Time to Progression（TTP）according to RECIST V1.1 criteria | From date of randomization until the date of first documented progression, up to 48 months
  efficacy
Time to Progression（TTP）according to mRECIST criteria | From date of randomization until the date of first documented progression, up to 48 months
  efficacy
Progresison Free Surviva（PFS）according to RECIST V1.1 criteria | From date of randomization until the date of the first documented progression or date of death from any cause, whichever comes first, up to 48 months
  efficacy
Progresison Free Surviva（PFS）according to mRECIST criteria | From date of randomization until the date of the first documented progression or date of death from any cause, whichever comes first, up to 48 months
  efficacy
Overall survival (OS) | From date of randomization until death from any cause，through study completion, an average of 3 years
  efficacy
Immune Best Overall Response（iBOR）according to iRECIST criteria | The best timepoint response recorded from the start of the study treatment until the end of treatment, taking into account any requirement for confirmation, through study completion, an average of 3 years
  efficacy